CLINICAL TRIAL: NCT03795220
Title: Preparing and Timing of the Endometrium in Modified Natural Cycle Frozen-thawed Embryo Transfers (mNC-FET) - a Randomized Controlled Multicenter Trial
Brief Title: Preparing and Timing of the Endometrium in Modified Natural Cycle Frozen-thawed Embryo Transfers
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Anja Bisgaard Pinborg (Other)
Collaborators: Copenhagen University Hospital, Hvidovre (Other); Regionshospitalet Horsens (Other); Copenhagen University Hospital at Herlev (Other); Aalborg University Hospital (Other); Hillerod Hospital, Denmark (Other); Zealand University Hospital (Other); Regionshospitalet Viborg, Skive (Other)
Responsible Party: Sponsor-Investigator, Anja Bisgaard Pinborg, Professor, chief consultant, DMSC, Rigshospitalet, Denmark
Organization: Rigshospitalet, Denmark (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 63569; 2018-002207-34 (EudraCT Number)
Record Dates: First submitted 2018-12-04; First posted 2019-01-07 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2024-02

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility

STUDY DESIGN:
Intervention Model Description: Randomized, controlled multicenter trial with inclusion of 604 mNC-FET cycles. We will include 604 patients divided 1:1 (302:302) in each arm +/- progesterone supplementation and these will further be divided 1:1 in blastocyst warming and transfer +6 and +7 days after hCG injection. Patients randomised to progesterone supplementation will start administering medicine four days after the ovulation trigger up til the day of the pregnancy test. If the pregnancy test is positive, medication will continue for 30 days more.
Who Masked: Investigator
Masking Description: The study is a single blinded study; therefore, the study medication will be blinded for the treating doctors, but not for the patients, the non-treating doctors or the study nurses. Patients will only be seen by a treating doctor at the day of blastocyst transfer and at the day of the pregnancy scan. The participants will not take progesterone the morning of the blastocyst transfer, but immediately after to keep the treating doctors blinded. Patients will be instructed in not disclosing their study group to the treating doctor.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (4):
- Vaginal progesterone + transfer 6. day (Active Comparator): Lutinus + blastocyst warming and transfer 6 days after hCG trigger
  Interventions: Drug: Lutinus + transfer day 6
- Vaginal progesterone + transfer 7. day (Active Comparator): Lutinus + blastocyst warming and transfer 7 days after hCG trigger
  Interventions: Drug: Lutinus + transfer day 7
- No progesterone + transfer 6. day (Active Comparator): No Lutinus + blastocyst warming and transfer 6 days after hCG trigger
  Interventions: Drug: No Lutinus + transfer day 6
- No progesterone + transfer 7. day (Active Comparator): No Lutinus + blastocyst warming and transfer 7 days after hCG trigger
  Interventions: Drug: No Lutinus + transfer day 7

INTERVENTIONS:
Drug: Lutinus + transfer day 6 — Four parallel groups of patients undergoing fertility treatment (modified natural cycle frozen embryo transfer) will be compared using/not using vaginal progesterone (Lutinus) and subject to blastocyst warming and transfer 6/7 days after hCG trigger.
  Other Names: Lutinus
  Arms: Vaginal progesterone + transfer 6. day
Drug: Lutinus + transfer day 7 — Four parallel groups of patients undergoing fertility treatment (modified natural cycle frozen embryo transfer) will be compared using/not using vaginal progesterone (Lutinus) and subject to blastocyst warming and transfer 6/7 days after hCG trigger.
  Other Names: Lutinus
  Arms: Vaginal progesterone + transfer 7. day
Drug: No Lutinus + transfer day 6 — Four parallel groups of patients undergoing fertility treatment (modified natural cycle frozen embryo transfer) will be compared using/not using vaginal progesterone (Lutinus) and subject to blastocyst warming and transfer 6/7 days after hCG trigger.
  Arms: No progesterone + transfer 6. day
Drug: No Lutinus + transfer day 7 — Four parallel groups of patients undergoing fertility treatment (modified natural cycle frozen embryo transfer) will be compared using/not using vaginal progesterone (Lutinus) and subject to blastocyst warming and transfer 6/7 days after hCG trigger.
  Arms: No progesterone + transfer 7. day

SUMMARY:
The increasing use of FET emphasizes the importance of preparing and timing the endometrium in FET cycles, however there is no consensus on luteal phase progesterone supplementation in mNC-FET and the optimal day of blastocyst warming and transfer. The aim of this multicenter RCT is to assess the effect of progesterone supplementation in hCG-triggered mNC-FET and the effect of embryo thawing and transfer at hCG+6 or hCG+7 days, respectively. In total 604 patients will be included with n=151 in each of the four study arms. The primary outcome is live birth rate per transfer (LBR) and the goal is to show a 10% increase in LBR after progesterone supplementation and to assess whether blastocyst warming+transfer 6 days after hCG trigger is superior to 7 days after hCG trigger in mNC-FET.

DETAILED DESCRIPTION:
Single embryo transfer and freezing of surplus embryos has lowered twin birth rates after in vitro fertilization (IVF) to a level of less than 5% in Denmark. However, several treatments with repeated frozen embryo transfers (FET) before a viable pregnancy is confirmed are burdensome to the patients. New freezing techniques has optimized the quality of the embryo transferred in FET cycles, but optimization of the endometrium in the luteal phase is still lacking behind. In a mNC-FET, which is the routine in many clinics, ovulation is induced with an hCG injection when the leading follicle is ≥17 mm. The hCG trigger is important for controlling the time of ovulation, but triggering an unhealthy follicle at an inappropriate time may cause luteal phase insufficiency and thus suboptimal function of the endometrium. Danish public fertility clinics are not routinely using progesterone supplementation in mNC-FET, but there may be a rationale to do so, and some implantations may be rescued. In this study we will compare live birth rates in mNC-FET with and without progesterone supplementation in the luteal phase, and further we will explore the optimal timing of blastocyst warming and transfer by comparing embryo transfer at hCG trigger +6 days versus +7 days. This is a superiority study with the aim to detect an increase in live birth rates of 10%. Hence, this adequately powered RCT may make a major contribution to knowledge on mNC-FET to the benefits of patients. We will include 604 patients divided 1:1 (302:302) in each arm +/- progesterone and these will further be divided 1:1 in blastocyst warming and transfer +6 and +7 days after hCG injection. The primary endpoint is live birth rate per transfer.

ELIGIBILITY:
Inclusion Criteria:

* Female age 18-41 years, regular menstrual cycle (23-35 days), vitrified blastocysts derived from 1.-3. IVF/ICSI cycle in a public hospital and undergoing single blastocyst transfer.

Exclusion Criteria:

- Previous participation in the study, uterine malformations, intrauterine polyps or submucosal myomas, breast feeding, oocyte donation, preimplantation genetic testing, blastocyst conceived with sperm from testicular sperm aspiration, HIV (woman), hepatitis B and C (woman), known luteal phase insufficiency or if patients are not fulfilling the inclusion criteria. Further exclusion criteria are the following contraindications to progesterone; allergy to the study medication, undiagnosed vaginal bleeding, current missed abortion or ectopic pregnancy, hepatic insufficiency or severe hepatic disease, genital or breast cancer, arterial or venous thromboembolism, thrombophlebitis or porphyria. For patients participating in the sub-study, thyroid disease is an exclusion criterion.

Ages: 18 Years to 41 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 679 (Actual)
Dates: Start 2019-01-06 (Actual); Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Live birth rates per transfer | Registered at the one-year follow-up after a positive pregnancy test.
  Comparison of live birth rates between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.

SECONDARY OUTCOMES:
Chemical pregnancy rates per transfer | Measured 16 days after ovulation trigger (hCG+16).
  Comparison of chemical pregnancy rates between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Clinical pregnancy rates per transfer | Ultrasound performed at 7-8 weeks of gestation.
  Comparison of clinical pregnancy rates (ultrasound) between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or seven after hCG trigger.
Abortion rates per transfer | Registered at the one-year follow-up after a positive pregnancy test.
  Comparison of abortion rates between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
ASAT (U/L) | Measured at baseline.
  ALAT measured by blood sample to ensure normal liver parameters before administration of progesterone.
ALAT (U/L) | Measured at baseline.
  ALAT measured by blood sample to ensure normal liver parameters before administration of progesterone.
AMH (pol/L) | Measured at baseline.
  Comparison of AMH measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Estradiole (mmol/L) | Measured at baseline, at ovulation trigger day (hCG+0), at transfer day (hCG+6/7) and at hCG+11.
  Comparison of estradiole measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
FSH (IU/L) | Measured at baseline, at ovulation trigger day (hCG+0), at transfer day (hCG+6/7) and at hCG+11.
  Comparison of FSH measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
LH (IU/L) | Measured at baseline, at ovulation trigger day (hCG+0), at transfer day (hCG+6/7) and at hCG+11.
  Comparison of LH measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Progesterone (nmol/L) | Measured at baseline, at ovulation trigger day (hCG+0), at transfer day (hCG+6/7) and at hCG+11.
  Comparison of progesterone measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
OH-progesterone (nmol/L) | Measured at ovulation trigger day (hCG+0), at transfer day (hCG+6/7) and at hCG+11.
  Comparison OH-progesterone measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
beta-hCG | Measured at transfer day (hCG+6/7), hCG+11 and hCG+16.
  Comparison of beta-hCG measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
TSH (*10^3 IU/L) | Measured at baseline, at ovulation trigger day (hCG+0), at transfer day (hCG+6/7), at hCG+11, at hCG+14 and at hCG+19.
  Comparison of TSH measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Thyroglobulin antibodies (arb.units/L) | Measured at baseline.
  Comparison of thyroglobulin antibodies measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Thyroid peroxidase anitbodies (arb.units/L) | Measured at baseline.
  Comparison of thyroid peroxidase antibodies measured by blood samples between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Obstetric complication rates | Registered at the one-year follow-up after a positive pregnancy test.
  Comparison of obstetric complication rates between patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.
Neonatal complication rates | Registered at the one-year follow-up after a positive pregnancy test.
  Comparison of neonatal complication rates for children of patients receiving and not receiving Lutinus, with blastocyst warming and transfer day 6 or 7 after hCG trigger.

CONTACTS AND LOCATIONS:
Overall Officials: Anja B. Pinborg, Prof., DMSC, Principal Investigator — Rigshospitalet, Denmark
Locations (1):
- Fertility Clinic, Rigshospitalet, Copenhagen University Hospital, Copenhagen, Denmark

IPD SHARING:
Plan to Share IPD: Yes
On request the study protocol and deidentified individual study data collected during the trial, including stored biobank samples, can be shared with research groups with relevant aims and a methodologically sound proposal. Approvals by necessary ethic committees and the Danish Data Protection Agency will be needed before sharing of data. All costs for data sharing will be covered by the party requesting the data. Data cannot be shared with groups working on research projects with the same aims, secondary aims or purposes. Further no data can be shared until 3 months after publication of first papers on the primary and secondary outcomes in this study. Biobank samples cannot be shared with research groups outside Denmark. Proposals of data sharing should be directed to anja.bisgaard.pinborg@regionh.dk. To gain access, data requestors will need to sign a data sharing agreement.
Supporting Information: Study Protocol
Time Frame: Data will be available from 3 months after publication of first papers on the primary and secondary outcomes in this study.
Access Criteria: Approvals by necessary relevant ethic committees and the Danish Data Protection Agency will be needed before sharing of data. All costs for data sharing will be covered by the party requesting the data. Data cannot be shared with groups working on research projects with the same aims, secondary aims or purposes. Biobank samples cannot be shared with research groups outside Denmark.

REFERENCES:
- [Derived] Saupstad M, Colombo C, Bergenheim SJ, Pistoljevic-Kristiansen N, Dam TV, Bogstad JW, Praetorius L, Freiesleben NC, Klajnbard A, Oxlund-Mariegaard B, Humaidan P, Lokkegaard ECL, Husth M, Knudsen UB, Gabrielsen A, Forman JL, Petersen MR, Lossl K, Pinborg A. Optimizing the protocol for modified natural cycle frozen embryo transfer (mNC-FET): a multicentre, single-blinded randomized controlled trial. Hum Reprod Open. 2026 Jan 13;2026(1):hoag003. doi: 10.1093/hropen/hoag003. eCollection 2026. PMID 41640422
- [Derived] Colombo C, Pistoljevic-Kristiansen N, Saupstad M, Bergenheim SJ, Spangmose AL, Klajnbard A, la Cour Freiesleben N, Lokkegaard EC, Englund AL, Husth M, Breth Knudsen U, Alsbjerg B, Praetorius L, Lossl K, Schmidt L, Pinborg A. Does luteal phase progesterone supplementation affect physical and psychosocial well-being among women undergoing modified natural cycle-FET? A sub-study of a randomized controlled trial. Hum Reprod. 2023 Oct 3;38(10):1970-1980. doi: 10.1093/humrep/dead171. PMID 37634089
- [Derived] Saupstad M, Freiesleben NC, Skouby SO, Andersen LF, Knudsen UB, Petersen KB, Husth M, Egeberg A, Petersen MR, Ziebe S, Andersen AN, Lossl K, Pinborg A. Preparation of the endometrium and timing of blastocyst transfer in modified natural cycle frozen-thawed embryo transfers (mNC-FET): a study protocol for a randomised controlled multicentre trial. BMJ Open. 2019 Dec 15;9(12):e031811. doi: 10.1136/bmjopen-2019-031811. PMID 31843833